CLINICAL TRIAL: NCT05825963
Title: Enrichment of Hamburger Meatballs With Psyllium and Determination of the Effects on Postprandial Lipidemia, Glycemia, Appetite, and Food Intake
Brief Title: Psyllium-enriched Hamburger Meatballs: Effects on Postprandial Lipidemia, Glycemia, Appetite, and Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmet Murat Günal (Other)
Responsible Party: Sponsor-Investigator, Ahmet Murat Günal, Assistant Professor Doctor, Okan University
Organization: Okan University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IstanbulOkanU
Record Dates: First submitted 2023-03-24; First posted 2023-04-24 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Nutrition, Healthy; Appetitive Behavior; Food Preferences; Obesity; Cardiovascular Diseases
Keywords: Psyllium; soluble fiber; hamburger; postprandial lipidemia; food intake; appetite
MeSH Terms: conditions — Appetitive Behavior; Food Preferences; Obesity; Cardiovascular Diseases | interventions — Psyllium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEHM/CHM (Experimental): In this arm, participants received psyllium-enriched hamburger meatballs first, then after the washout period, they received classic hamburger meatballs.
  Interventions: Dietary Supplement: Psyllium
- CHM/PEHM (Experimental): In this arm, participants received classic hamburger meatballs first, then after the washout period, they received psyllium-enriched hamburger meatballs.
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Dietary Supplement: Psyllium — The participants select hamburgers randomly by themselves, with or without (control) 12 g of psyllium, each containing 85 g of hamburger bread, 160 g of 20% fat beef, 2.56 g of salt, and 1.28 g of pepper, and asked to consume them with 200 ml of water.

SUMMARY:
The goal of this clinical trial is to enrich the hamburger meatball with psyllium without impairing its sensory properties and to investigate the effects on acute postprandial lipemia and glycemia, prospective food intake, and some appetite indicators in healthy adults. The main hypotheses of the study are:

1. There is no difference in sensory analysis results between hamburger meatballs enriched with psyllium and those that are not enriched.
2. The rise in postprandial lipids after consuming psyllium-enriched hamburger meatballs is lower than that of classic hamburgers.
3. The rise in postprandial glycemia after consuming psyllium-enriched hamburger meatballs is lower than that of classic hamburgers.
4. The feeling of satiety after consuming psyllium-enriched hamburger meatballs lasts longer, and the feeling of hunger lasts for a shorter period compared to classic hamburgers.
5. Daily food intake after consuming psyllium-enriched hamburger meatballs is less than that of classic hamburgers.

Participants will,

* Eat hamburgers, after fasting for 12 hours, with psyllium-enriched and classic meatballs on intervention days.
* Keep a record of their food intake for the previous and following 24 hours of each intervention.
* Be given fasting and postprandial blood samples.
* Evaluate their hunger and satiety levels on a 100 mm horizontal visual analog scale (VAS) at the beginning and every hour for the following 6 hours of the study.

DETAILED DESCRIPTION:
After preparing 7.5% psyllium-enriched hamburger meatballs (PEHMs) and control hamburger meatballs (CHMs), they will be placed in identical storage containers and frozen at -18°C in a deep freezer. An independent academic will use the Google Random Number Generator to randomly assign two three-digit numbers and code each group accordingly to ensure that the experimental period will be triple-blind.

Participants will be asked to keep a record of their food intake for the previous 24 hours, avoid heavy physical activity, abstain from alcohol before the first day of the study, and to arrive at the study in a state of fasting for 12 hours. On the study day, the participants' sociodemographic information will be collected, anthropometric measurements (height, weight, and fat percentage) will be taken, and fasting blood samples will be collected by a nurse. The participants will then select hamburgers randomly by themselves, with or without (control) 12 g of psyllium, each containing 85 g of hamburger bread, 160 g of 20% fat beef, 2.56 g of salt, and 1.28 g of pepper. They will be asked to consume them with 200 ml of water. The codes for the hamburgers will be written under the plate. The researcher will record which participant consumed which coded hamburger. After waiting two hours in a designated room, postprandial blood samples will be collected in the same order and sent for analysis.

After analyzing the fasting blood values of the participants, if any of them have dyslipidemia (LDL> 149) will be excluded from the study. The remaining participants will be invited back for the second day of the study following a two-week washout period. On this day, the hamburger that they did not consume on the first day will be served to them and the same procedure will repeat.

The guidelines outlined in the CONSORT 2010 statement will be followed during the conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being willing to participate in the research
* Aged 19 to 35
* No chronic or metabolic disorders
* Body mass index (BMI) between 18.5 and 25 kg/m2

Exclusion Criteria:

* Not being willing to participate in the research,
* Having chronic diseases such as diabetes, hypertension, cancer, metabolic syndrome, chronic kidney disease, dyslipidemia, etc.
* Having a congenital metabolic disease,
* Taking medication to lower blood lipids,
* Being pregnant or breastfeeding,
* Being vegan or vegetarian (as the study requires meat consumption).

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-08-17 (Actual)

PRIMARY OUTCOMES:
Postprandial changes in lipid profile | 0 and 2nd hours of each intervention
  Comparison of participants' fasting and postprandial lipid levels according to the hamburgers consumed (mg/dL) will be conducted.
Postprandial changes in glycemia | 0 and 2nd hours of each intervention
  Comparison of participants' fasting and postprandial glucose levels according to the hamburgers consumed (mg/dL) will be conducted.
Postprandial changes in satiety and hunger | Change from baseline to 6th hours of each intervention
  Comparison of participants' subjective evaluations of hunger and satiety according to the hamburgers consumed will be conducted using visual analog scale (VAS). Which is a 100mm horizontal scale, indicating stronger feelings (satiety, hunger) toward 100.
Changes in daily food intake | Change from one day before to one day after of each intervention
  Comparison of participants' food intake according to the hamburgers consumed will be conducted using 24-hour food intake record.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Murat Günal, Ph.D., Principal Investigator — Okan University
Locations (1):
- İstanbul Okan University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPDs will be shared after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 mounts after publication
Access Criteria: For systematic review and meta-analyses.

REFERENCES:
- [Background] Phan JL, Cowley JM, Neumann KA, Herliana L, O'Donovan LA, Burton RA. The novel features of Plantago ovata seed mucilage accumulation, storage and release. Sci Rep. 2020 Jul 16;10(1):11766. doi: 10.1038/s41598-020-68685-w. PMID 32678191
- [Background] Fischer MH, Yu N, Gray GR, Ralph J, Anderson L, Marlett JA. The gel-forming polysaccharide of psyllium husk (Plantago ovata Forsk). Carbohydr Res. 2004 Aug 2;339(11):2009-17. doi: 10.1016/j.carres.2004.05.023. PMID 15261594
- [Background] Gibb RD, McRorie JW Jr, Russell DA, Hasselblad V, D'Alessio DA. Psyllium fiber improves glycemic control proportional to loss of glycemic control: a meta-analysis of data in euglycemic subjects, patients at risk of type 2 diabetes mellitus, and patients being treated for type 2 diabetes mellitus. Am J Clin Nutr. 2015 Dec;102(6):1604-14. doi: 10.3945/ajcn.115.106989. Epub 2015 Nov 11. PMID 26561625
- [Background] McRorie JW Jr. Evidence-Based Approach to Fiber Supplements and Clinically Meaningful Health Benefits, Part 1: What to Look for and How to Recommend an Effective Fiber Therapy. Nutr Today. 2015 Mar;50(2):82-89. doi: 10.1097/NT.0000000000000082. PMID 25972618
- [Background] Wanders AJ, van den Borne JJ, de Graaf C, Hulshof T, Jonathan MC, Kristensen M, Mars M, Schols HA, Feskens EJ. Effects of dietary fibre on subjective appetite, energy intake and body weight: a systematic review of randomized controlled trials. Obes Rev. 2011 Sep;12(9):724-39. doi: 10.1111/j.1467-789X.2011.00895.x. Epub 2011 Jun 16. PMID 21676152
- [Background] Howarth NC, Saltzman E, Roberts SB. Dietary fiber and weight regulation. Nutr Rev. 2001 May;59(5):129-39. doi: 10.1111/j.1753-4887.2001.tb07001.x. PMID 11396693
- [Background] Trumbo P, Schlicker S, Yates AA, Poos M; Food and Nutrition Board of the Institute of Medicine, The National Academies. Dietary reference intakes for energy, carbohydrate, fiber, fat, fatty acids, cholesterol, protein and amino acids. J Am Diet Assoc. 2002 Nov;102(11):1621-30. doi: 10.1016/s0002-8223(02)90346-9. No abstract available. PMID 12449285
- [Background] Isganaitis E, Lustig RH. Fast food, central nervous system insulin resistance, and obesity. Arterioscler Thromb Vasc Biol. 2005 Dec;25(12):2451-62. doi: 10.1161/01.ATV.0000186208.06964.91. Epub 2005 Sep 15. PMID 16166564
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Khossousi A, Binns CW, Dhaliwal SS, Pal S. The acute effects of psyllium on postprandial lipaemia and thermogenesis in overweight and obese men. Br J Nutr. 2008 May;99(5):1068-75. doi: 10.1017/S0007114507864804. Epub 2007 Nov 16. PMID 18005484
- [Background] Pal S, Ho S, Gahler RJ, Wood S. Effect on Insulin, Glucose and Lipids in Overweight/Obese Australian Adults of 12 Months Consumption of Two Different Fibre Supplements in a Randomised Trial. Nutrients. 2017 Jan 29;9(2):91. doi: 10.3390/nu9020091. PMID 28146065
- [Background] Brennan MA, Derbyshire EJ, Brennan CS, Tiwari BK. Impact of dietary fibre-enriched ready-to-eat extruded snacks on the postprandial glycaemic response of non-diabetic patients. Mol Nutr Food Res. 2012 May;56(5):834-7. doi: 10.1002/mnfr.201100760. PMID 22648629
- [Background] Pal S, Khossousi A, Binns C, Dhaliwal S, Ellis V. The effect of a fibre supplement compared to a healthy diet on body composition, lipids, glucose, insulin and other metabolic syndrome risk factors in overweight and obese individuals. Br J Nutr. 2011 Jan;105(1):90-100. doi: 10.1017/S0007114510003132. Epub 2010 Aug 23. PMID 20727237
- [Background] Karhunen LJ, Juvonen KR, Flander SM, Liukkonen KH, Lahteenmaki L, Siloaho M, Laaksonen DE, Herzig KH, Uusitupa MI, Poutanen KS. A psyllium fiber-enriched meal strongly attenuates postprandial gastrointestinal peptide release in healthy young adults. J Nutr. 2010 Apr;140(4):737-44. doi: 10.3945/jn.109.115436. Epub 2010 Feb 10. PMID 20147463
- [Background] Brum JM, Gibb RD, Peters JC, Mattes RD. Satiety effects of psyllium in healthy volunteers. Appetite. 2016 Oct 1;105:27-36. doi: 10.1016/j.appet.2016.04.041. Epub 2016 May 7. PMID 27166077
- [Derived] Gunal AM, Ongun Yilmaz H, Bas M. Enrichment of Hamburger Meatballs With Psyllium: Effects on Postprandial Lipidemia, Glycemia, Appetite, and Food Intake in a Triple-Blind Randomized Controlled Crossover Trial. Food Sci Nutr. 2025 Oct 9;13(10):e71066. doi: 10.1002/fsn3.71066. eCollection 2025 Oct. PMID 41078451